CLINICAL TRIAL: NCT03751046
Title: Controlled Clinical Trial Comparing the Efficacy of Trial-Based Cognitive Therapy and Standard Care for the Treatment of HIV+ Patients With Antiretroviral Therapy Failure, Bogotá, Colombia
Brief Title: Cognitive Therapy in Patients Failing ART
Acronym: CognitiveTher
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundação Bahiana de Infectologia (Other)
Responsible Party: Principal Investigator, Monica Bibiana Narvaez Betancur, Principal investigator, Fundação Bahiana de Infectologia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EC003; U1111-1219-0997 (Other: IRB Bogotá)
Record Dates: First submitted 2018-11-09; First posted 2018-11-23 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: HIV; Cognitive Therapy
Keywords: HIV; Cognitive therapy; Treatment; HAART; Treatment adherence and compliance
MeSH Terms: conditions — Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group. Trial-Based Cognitive Therapy (Experimental): Participants with therapeutic failure. Fourteen sessions of psychotherapy in group format, using Trial-Based Cognitive Therapy. Frequency: Bi-weekly meetings for seven months. Intervention arm comprises 10 psychotherapy groups with five participants in each group.
  Interventions: Behavioral: Trial-Based Cognitive Therapy
- Control group. Standard healthcare. (Experimental): Participants with therapeutic failure, receiving standard healthcare in the HIV/AIDS Program, which includes at least half-yearly psychology and pharmaceutical chemist consultations (approximately half an hour each). The purpose of these consultations is to approach the importance of adherence and psychoeducation on HIV.
  Interventions: Other: Control group. Standard healthcare.

INTERVENTIONS:
Behavioral: Trial-Based Cognitive Therapy — Participants in the TBCT intervention arm will have 14 (fourteen) psychotherapy sessions over a period of 7 (seven) months. The frequency of the intervention is biweekly with a duration of approximately 90 minutes per session. We will have10 groups with 5 participants each. All participants will practice the learned techniques during the meetings, have a manual with a description summary of the sessions and the activities to practice at home. The main TBCT techniques that will be used are case conceptualization, intrapersonal thought record, consensual role-play, action plan, trial-based thought record and trial-based metacognitive awareness.
  Other Names: TBCT
  Arms: Intervention group. Trial-Based Cognitive Therapy
Other: Control group. Standard healthcare. — Participants with therapeutic failure, receiving the standard healthcare in the HIV / AIDS Program, which includes at least a half-yearly psychology and pharmaceutical chemist consultations (approximately half an hour each).
  The purpose of these consultations is to approach the importance of adherence and psychoeducation on HIV
  Other Names: Standard healthcare
  Arms: Control group. Standard healthcare.

SUMMARY:
Highly active antiretroviral therapy (HAART) has been the greatest achievement to control the HIV/AIDS epidemic in the world. HAART has been shown to reduce virus replication to undetectable levels and to favor the recovery of immune function, avoiding the occurrence of opportunistic diseases. Although existing treatments have been shown to lower AIDS-related morbimortality and to increase patients' quality of life, the success of HAART requires high levels of adherence to the prescribed treatment regimen.

Adherence to HAART has become the major challenge for global public policy managers and healthcare teams involved in the care of HIV/AIDS patients. Mental healthcare professionals should use structured and effective intervention as strategies to facilitate a better approach, increase patients' autonomy and achieve optimal adherence.

Trial-Based Cognitive Therapy (TBCT) is a new, structured, and short-term version of cognitive behavior therapy developed by de Oliveira (2011). TBCT is an active approach that aims to change negative cognitions, especially dysfunctional core beliefs, that negatively influence patient's life in different domains. TBCT helps patients recognize situationally based thoughts, unhelpful beliefs and maladaptive behaviors that exacerbate emotional distress.

This study aims to assess the efficacy of TBCT in helping the patients to identify thoughts, emotions, assumptions and behaviors associated with non-adherence to antiretroviral therapy, and to improve adherence to treatment.

ELIGIBILITY:
Inclusion Criteria:

* The last two detectable CV > 500 copies
* At least one year of antiretroviral treatment
* Age between 18 and 65 years
* Literate person.

Exclusion Criteria:

* Difficulty to read and to write
* Being currently in psychotherapy
* Clinical diagnoses of neurocognitive or psychotic disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-03-17 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
Change in adherence levels to antiretroviral treatment | Baseline, seven, ten and thirteen months after the baseline
  The primary efficacy measure is the improvement in adherence to antiretroviral therapy, measured by self-registration of adherence follow-up questionnaire (QOL 702) ACTG (the Clinical Trials Group). This questionnaire assesses the percentage of self-reported adherence in the last 4 days and the reasons for not taking medicines. Individuals who take 95% or more of the prescribed doses are considered adherent. The analyses will be carried out comparing baseline measures with those observed as at seven, ten and thirteen months after the baseline measures in each group; also, comparisons between the intervention group and the control group will be carried out.

SECONDARY OUTCOMES:
Change in HIV-1 Viral Load | Baseline, seven, ten and thirteen months after the baseline
  Change in the number of copies in the HIV-1 Viral Load laboratory test result to <50 copies. The analyses will be carried out comparing the results in the baseline times, the results evaluated as at seven, ten and thirteen months after the baseline measures in each group and the comparison between the intervention group and the control group.
Change in depression levels | Baseline, seven, ten and thirteen months after the baseline
  Change in depression levels measured by the Beck Depression Inventory (BDI-II), which ranks in four levels according to the following scores: minimum (0-13), moderate (14-19), mild (20-28) and severe (29-63).The analyses will be carried out comparing baseline measures with those observed as at seven, ten and thirteen months after the baseline measures in each group and the comparison between the intervention group and the control group.
Changing anxiety levels | Baseline, seven, ten and thirteen months after the baseline
  Change in anxiety levels measured by the Beck Inventory for Anxiety (BAI), which ranks in four levels according to scores: minimum (0-7), moderate (8-15), mild (16-25), and severe (26-63).The analyses will be carried out comparing baseline measures with those observed as at seven, ten and thirteen months after the baseline measures in each group and the comparison between the intervention group and the control group.
Change in health-related quality of life measured by The Short Form Health Survey questionnaire , SF36 | Baseline, seven, ten and thirteen months after the baseline
  The instrument comprises eight multi-item scales: physical functioning, role limitations due to physical problems, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems and mental health. The eight multi-item scales are aggregated into a physical component (PCS) and a mental component summary (MCS) score.
  Physical functioning, role limitations due to physical problems, and bodily pain contribute more significantly to the PCS.
  Social functioning, role limitations due to emotional problems, and mental health contribute more significantly to MCS.
  The normalized scoring of the eight scales using the original 0 to 100 algorithms (raw scores) and the two summary components is performed by OPTUM PRO CoRETM Scoring Software based on norms with a mean of 50 and a standard deviation of 10. Normalized scores allow comparison of the eight domains and quantification of the SF-36 domains that are most affected by specific risk factors.
Change in health-related quality of life measured by WHOQOL-VIH BREF | Baseline, seven, ten and thirteen months after the baseline
  The instrument has 31 items with some specific items related to HIV/AIDS. Individual items are rated on a 5 point Likert scale where 1 indicates low, negative perceptions and 5 indicates high, positive perceptions. The instrument is scored in six domains: physical health; psychological health; level of independence; social relationship; environmental health and spirituality.
  Domain and facet scores are scaled in a positive direction where higher scores denote higher quality of life. Some facets (Pain and Discomfort, Negative Feelings, Dependence on Medication, Death and Dying) are not scaled in a positive direction, meaning that for these facets higher scores do not denote higher quality of life. These need to be recoded so that high scores reflect better QoL.
  Items are organised by response scale (capacity, frequency, intensity or satisfaction). Instructions for calculation of scores,using the original 0 to 100 algorithms, was obtained from the WHOQOL HIV Coordinator.

CONTACTS AND LOCATIONS:
Overall Officials: Mónica B Narváez, Psychologist, Master, Principal Investigator — Federal University of Bahia; Carlos R Brites, Post-Doctoral, Study Chair — Federal University of Bahia
Locations (1):
- Liga Colombiana de Lucha Contra El Sida, Bogotá, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No